CLINICAL TRIAL: NCT07006571
Title: Evaluation of the Efficacy of Home-based Transcranial Direct Current Stimulation on Physical Function in Patients With Amyotrophic Lateral Sclerosis: a Randomized, Controlled Clinical Trial
Brief Title: At-home Treatment With Cortico-spinal tDCS for Amyotrophic Lateral Sclerosis
Acronym: tDCS-ALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Alberto Benussi, Professor, University of Trieste
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 371/2024H
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: ALS; ALS (Amyotrophic Lateral Sclerosis)
Keywords: At-home tDCS; ALS; tDCS-ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS (Experimental): The device used for transcranial direct current stimulation (tDCS) is the Soterix Medical 1x1 tES mini-CT. The device is designed to be used at home by patients, with built-in safety controls to ensure adequate and safe stimulation. The electrodes of the device will be positioned according to the following scheme: one electrode (anode) will be applied on the skin overlying the motor cortices, one electrode (cathode) will be applied on the skin overlying the cervical cord, in the area corresponding to C6. Dosage: 4 mA for the anodal electrode and 4 mA for the cathodal electrode (intensity could be reduced if not tollerate by the patient).
  Duration of stimulation: 20 minutes per session. Frequency: 5 days per week (Monday - Friday) for 16 weeks.
  Interventions: Device: Real tDCS
- Sham tDCS (Sham Comparator): The placebo device uses the same model as the tDCS device but without actually delivering the current. The electrodes will be positioned in the same way as the active device, but the current flow will be limited to the ramp-up (start of stimulation) and ramp-down (end of stimulation) phase, mimicking the sensation of stimulation without providing actual treatment.
  Dosage: Simulation of stimulation without actual current. Duration of stimulation: 20 minutes per session. Frequency: 5 days per week (Monday - Friday) for 16 weeks.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Real tDCS — The electrodes of the device will be positioned according to the following scheme: one electrode (anode) will be applied on the skin overlying the motor cortices, one electrode (cathode) will be applied on the skin overlying the cervical cord, in the area corresponding to C6. Dosage: 4 mA for the anodal electrode and 4 mA for the cathodal electrode (intensity could be reduced if not tollerate by the patient). Duration of stimulation: 20 minutes per session. Frequency: 5 days per week (Monday - Friday) for 16 weeks.
  Arms: Real tDCS
Device: Sham tDCS — The electrodes will be positioned in the same way as the active device, but the current flow will be limited to the ramp-up (start of stimulation) and ramp-down (end of stimulation) phase, mimicking the sensation of stimulation without providing actual treatment. Dosage: Simulation of stimulation without actual current. Duration of stimulation: 20 minutes per session. Frequency: 5 days per week (Monday - Friday) for 16 weeks.
  Arms: Sham tDCS

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a progressive neurological disease that causes gradual muscle weakness and loss of muscle mass. It affects all muscles that control movement, speech, swallowing, and breathing. Unfortunately, ALS is currently incurable, and treatments are limited. Only two medications, riluzole and edaravone, have been approved and can slightly extend survival, typically between 20 and 48 months from diagnosis.

Recent research has identified a useful biomarker known as neurofilament light chain (NfL), which increases in the blood as nerve cells become damaged. Measuring NfL levels can help track the progression of ALS.

A promising non-invasive treatment called transcranial direct current stimulation (tDCS) has shown potential benefits for patients with ALS. tDCS involves safely applying mild electrical currents to specific areas of the brain and spinal cord. This approach aims to stimulate nerve cells, potentially improving their function and slowing disease progression. Initial studies have reported temporary improvements in muscle strength and survival when tDCS was used over a short period.

Based on these encouraging results, our study proposes a new home-based tDCS treatment program specifically designed for ALS patients. Participants will use an easy-to-operate, safe, and portable device at home. The treatment involves placing electrodes on the scalp and the neck area to stimulate both the motor areas of the brain and the spinal cord. Therapy sessions will occur five days per week over 16 weeks.

This home-based approach allows patients to comfortably receive therapy without daily trips to the hospital, making treatment more accessible and convenient. By providing this therapy at home, the investigators aim to improve the quality of life for ALS patients and explore new possibilities in treating and managing ALS and other neurodegenerative diseases.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is an irreversible neurodegenerative disorder characterized by progressive muscle weakness and atrophy, affecting all skeletal and respiratory muscles. This leads to increasing difficulties in speech, swallowing, and ultimately breathing. A progressive rise in neurofilament light chain (NfL) levels-biomarkers of neuronal damage-has also been documented and may serve as a tool for monitoring disease progression. Average survival ranges from 20 to 48 months. Currently, there is no cure for ALS. Only two drugs, riluzole and edaravone, have demonstrated a modest extension of survival. In this context, transcranial direct current stimulation (tDCS) has emerged as a promising non-invasive neuromodulatory technique capable of modulating central nervous system excitability. Its popularity is growing due to its simplicity, low cost, and broad therapeutic potential across various neurodegenerative conditions. tDCS exerts long-lasting effects on synaptic plasticity in the motor cortex, primarily through modulation of NMDA receptors and GABAergic systems. Given that ALS involves irreversible degeneration of both upper and lower motor neurons in the motor cortex and spinal cord, tDCS may offer therapeutic benefit. Preliminary studies have shown transient improvements in muscle strength and survival following cortico-spinal tDCS administered over two weeks.

Building on these findings, a protocol is proposed for home-based tDCS treatment in ALS patients, consisting of multiple sessions aimed at achieving greater and more sustained effects. A brain stimulation device specifically designed for home use will be employed. This device incorporates safety features that monitor for improper usage.

The procedure involves applying an anodal stimulation over the motor cortex bilaterally and a cathodal stimulation over the cervical spinal cord. Stimulation sessions will be conducted five days per week over a 16-week period. Home-based tDCS offers a safe alternative to hospital-based treatment, eliminating the need for daily travel and allowing patients to undergo therapy in the comfort of their own homes. This approach represents a potentially significant innovation in ALS care-offering a non-invasive, safe, and accessible therapeutic option that may enhance quality of life and open new avenues for research in neurodegenerative disease management.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a probable, laboratory-supported diagnosis of ALS, or defined ALS according to current clinical criteria
* Age greater than 18 years
* Onset of disease ≤ 24 months
* Disease progression in the last 3 months
* A score ≥ 2 on the "respiratory failure" item on the ALS Functional Rating Scale Revised (ALSFRS-R)
* Treatment with riluzole or edaravone is permitted, provided it has been stable for at least 1 month prior to enrollment in the study, or no ALS-specific treatment
* Presence of a caregiver who can assist the patient and who has successfully completed the necessary training in the use of the device
* Signature of informed consent

Exclusion Criteria:

* People with fixed electrical stimulators (e.g. cardiac pacemakers, nerve stimulators, hearing implants) that would not work or would be damaged by the electric field;
* People with particular intracranial metal foreign bodies (e.g. splinters, some prostheses, screws and nails) that could interact with the electric field
* People with a history of epilepsy;
* As the effects of tDCS on the developing fetus are not known, pregnant women will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Difference in the ALSFRS-R between groups at 16 weeks. | Baseline - 16 weeks
  Difference in ALS Functional Rating Scale-Revised (ALSFRS-R) between groups at 16 weeks. The ALSFRS provides a physician-generated estimate of the patient's degree of functional impairment, which can be evaluated serially to objectively assess any response to treatment or progression of disease. The ALSFRS includes ten questions that rate the patients level of functional impairment in performing one of ten common tasks. Each task is rated on a five-point scale from 0 (can't do) to 4 (normal ability). Individual item scores are summed to produce a reported score of between 40 (no impairment) and 0 (severe impairment).

SECONDARY OUTCOMES:
Difference in the ALSFRS-R between groups at 32 weeks and 48 weeks | 32 weeks - 48 weeks
  Difference in the ALS Functional Rating Scale-Revised (ALSFRS-R) between groups at 32 weeks and 48 weeks. The ALSFRS provides a physician-generated estimate of the patient's degree of functional impairment, which can be evaluated serially to objectively assess any response to treatment or progression of disease. The ALSFRS includes ten questions that rate the patients level of functional impairment in performing one of ten common tasks. Each task is rated on a five-point scale from 0 (can't do) to 4 (normal ability). Individual item scores are summed to produce a reported score of between 40 (no impairment) and 0 (severe impairment).
Difference in the ALSAQ-40 between groups | Baseline - 16 weeks - 32 weeks - 48 weeks
  Difference in the Amyotrophic Lateral Sclerosis Assessment Questionnaire-40 score (ALSAQ-40) from baseline.The Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ) is a patient self-report health status scale. The ALSAQ is specifically used to measure the subjective well-being of patients with amyotrophic lateral sclerosis. There are 40 items/questions with 5 discrete scales: physical mobility (10 items), activities of daily living and independence (10 items), eating and drinking (3 items), communication (7 items), emotional reactions (10 items). Patients are asked to think about the difficulties they may have experienced during the last two weeks (e.g. I have found it difficult to feed myself). Patients are asked to indicate the frequency of each event by selecting one of 5 options (Likert scale):
  never/rarely/sometimes/often/always or cannot do at all. The total ranges from 0 (no impairment) to 160 (severe impairment).
Difference in the Caregiver Burden Inventory (CBI) score between groups | Baseline - 16 weeks - 32 weeks - 48 weeks
  Difference in the Caregiver Burden Inventory (CBI) score between groups from baseline.The CBI scale is 24- item scale designed to assess the experience of caregivers of older people. The multidimensional instrument assesses five domains of burden (time-dependence, developmental, physical, social, and emotional). Items are scored on a 4-point scale, ranging from "not at all descriptive" to "very descriptive". The scale ranges from 0 (no impairment) to 96 (severe impairment).
Difference in Quality of Life EQ-5D-5L Scale between groups | Baseline - 16 weeks - 32 weeks - 48 weeks
  Difference in Quality of Life EQ-5D-5L Scale between groups from baseline.The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The scale ranges from 5 (no impairment) to 25 (severe impairment).
Difference in Muscle strength assessed by manual dynamometer from baseline | Baseline - 16 weeks - 32 weeks - 48 weeks
  Muscle strength will be evaluated using a handheld dynamometer, a validated tool for objective measurement of isometric muscle force. Muscle groups typically involved in ALS will be assessed bilaterally using standardized testing positions. For each muscle group, participants will be instructed to perform a maximal voluntary isometric contraction against the dynamometer for approximately 3-5 seconds. Two trials will be performed per muscle, and the highest peak force (measured in Newtons) will be recorded. The sum of 10 muscles per side (20 overall) will be evaluated.
Difference in Plasma neurofilament levels between groups | Baseline - 16 weeks - 32 weeks - 48 weeks
  Difference in Plasma neurofilament levels between groups from baseline. Neurofilament light chain (NfL), a well-established biomarker of neuroaxonal injury, can be reliably quantified in plasma (pNfL) and has shown superior diagnostic accuracy in differentiating patients with amyotrophic lateral sclerosis (ALS) from those with ALS mimic syndromes. In addition, numerous studies have emphasized the prognostic value of both cerebrospinal (cNfL) and plasma (pNfL) NfL levels, reporting strong correlations with disease progression rate (DPR) and overall survival. Notably, early longitudinal investigations indicate that pNfL levels remain relatively stable over the disease course, underscoring their promise as biomarkers for monitoring therapeutic response.
Difference in Survival from the onset of symptoms between groups | Continuously - 48 weeks
  Difference in Survival from the onset of symptoms between groups. Survival is defined as the time from the symptom onset to death from any cause. Patients who are alive at the time of the last follow-up are censored at the date of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Benussi, MD, Principal Investigator — University of Trieste
Locations (1):
- Clinica Neurologica, Azienda Sanitaria Universitaria Giuliano Isontina, Trieste, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benussi A, Di Lorenzo F, Dell'Era V, Cosseddu M, Alberici A, Caratozzolo S, Cotelli MS, Micheli A, Rozzini L, Depari A, Flammini A, Ponzo V, Martorana A, Caltagirone C, Padovani A, Koch G, Borroni B. Transcranial magnetic stimulation distinguishes Alzheimer disease from frontotemporal dementia. Neurology. 2017 Aug 15;89(7):665-672. doi: 10.1212/WNL.0000000000004232. Epub 2017 Jul 26. PMID 28747446
- [Background] Benussi A, Koch G, Cotelli M, Padovani A, Borroni B. Cerebellar transcranial direct current stimulation in patients with ataxia: A double-blind, randomized, sham-controlled study. Mov Disord. 2015 Oct;30(12):1701-5. doi: 10.1002/mds.26356. Epub 2015 Aug 14. PMID 26274840